CLINICAL TRIAL: NCT00402753
Title: Physical Exercise to Improve Physical Performance and Health Related Quality of Life in Hematopoietic Stem Cell Transplantation Recipients
Brief Title: Ambulatory Physical Exercise Program in Hematopoietic Stem Cell Transplantation Recipients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Daniel Uebelhart MD, University Hospital Zurich
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: EK-519
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Cancer, Exercise, Health Related Quality of Life, PBSCT
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Physical exercise group: Combined supervised physical activity: Endurance and Resistive strength
  Interventions: Behavioral: Ambulatory Physical Exercise Program
- Group 2 (No Intervention): Usual care control group

INTERVENTIONS:
Behavioral: Ambulatory Physical Exercise Program — supervised exercise, 2 x / week
  Arms: Group 1

SUMMARY:
The proposed study in an inception cohort of patients with hematological malignancies treated with PBSCT is designed to evaluate the effects of a physical exercise intervention on muscular-skeletal, physical activity and quality of life outcomes.

DETAILED DESCRIPTION:
Peripheral Stem Cell Transplantation is a frequently used therapy option to increase survival in hematological and lymphatic malignancies. These malignancies and their treatment are associated with numerous physical and psychological symptoms and severe side effects. Physical exercise has been proposed as a promising strategy for the treatment of some of these physical and psychological complaints, and various exercise interventions are currently available after cancer treatment. To date, promising preliminary results concerning exercise programs in PBSCT recipients were published with limited sample size populations. Results of musculoskeletal outcomes in PBSCT recipients after cancer treatment are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Status after high-dose chemotherapy following Hematopoietic Stem Cell Transplantation
* Willing to enter a physical exercise program
* Good understanding of the German language
* Written informed consent

Exclusion Criteria:

* Uncontrolled cardiovascular disease and myocardial infarction in the previous six months
* Uncontrolled hypertension
* Uncontrolled thyroid disease
* Uncontrolled diabetes
* Diagnosis of depression before entering the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal performance | Baseline -3 months - 6 months
Knee extension strength | Baseline -3 months - 6 months
Grip Strength | Baseline -3 months - 6 months
6 minute walk test | Baseline -3 months - 6 months
15-meter walking speed | Baseline -3 months - 6 months
and Health Related Quality of Life: (Physical function subscale of the EORTC-QLQ-C30 questionnaire). | Baseline -3 months - 6 months

SECONDARY OUTCOMES:
Role-,cognitive-,emotional-,social-,symptom scales and the global health and quality of life scale of the EORTC-QLQ-C30 Health Related Quality of Life questionnaire. | Baseline -3 months - 6 months
Self-reported fatigue | Baseline -3 months - 6 months
Self-reported and objectively assessed physical activity | Baseline -3 months - 6 months
Whole body composition | Baseline -3 months - 6 months
Haemotological values: e.g Hemoglobin | Baseline -3 months - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil K Aaronson, PhD, Study Chair — Division of Psychosocial Research & Epidemiology, The Netherlands Cancer Institute, Amsterdam, The Netherlands.
Locations (4):
- Hogeschool Utrecht, University of Professional Education, Faculty of Health Care, Chair of Lifestyle and Health, Utrecht, Netherlands
- Switzerland (3):
  - Cantonal Hospital Münsterlingen, Münsterlingen
  - Cantonal Hospital St.Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

REFERENCES:
- [Background] Knols R, Aaronson NK, Uebelhart D, Fransen J, Aufdemkampe G. Physical exercise in cancer patients during and after medical treatment: a systematic review of randomized and controlled clinical trials. J Clin Oncol. 2005 Jun 1;23(16):3830-42. doi: 10.1200/JCO.2005.02.148. PMID 15923576
- [Background] Schmitz KH, Holtzman J, Courneya KS, Masse LC, Duval S, Kane R. Controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. Cancer Epidemiol Biomarkers Prev. 2005 Jul;14(7):1588-95. doi: 10.1158/1055-9965.EPI-04-0703. PMID 16030088
- [Background] Galvao DA, Newton RU. Review of exercise intervention studies in cancer patients. J Clin Oncol. 2005 Feb 1;23(4):899-909. doi: 10.1200/JCO.2005.06.085. PMID 15681536